CLINICAL TRIAL: NCT01715298
Title: A 12-week Multi-center, Randomized, Double-blind, Placebo Controlled Study to Assess the Efficacy and Safety of NVA237 in Stable COPD Patients
Brief Title: NVA237 BID Versus Placebo Twelve-week Efficacy Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CNVA237A2318
Record Dates: First submitted 2012-10-24; First posted 2012-10-26 (Estimated); Results first posted 2015-03-11 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Anticholinergic; Antimuscarinic; Chronic Obstructive Airway Disease; Chronic Obstructive Lung Disease; Chronic Obstructive Pulmonary Disease; COPD; LAMA; Lung Disease; Lung Diseases, Obstructive; Lung Function; Muscarinic receptor antagonist; Pulmonary Disease, Chronic Obstructive; Respiratory Tract Diseases
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases; Lung Diseases, Obstructive; Respiratory Tract Diseases | interventions — Glycopyrrolate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- NVA237 (Experimental): NVA237 will be inhaled from a single-dose dry powder inhaler for a period of 12 weeks
  Interventions: Drug: NVA237
- Placebo (Placebo Comparator): Placebo will be inhaled from a single-dose dry powder inhaler for a period of 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NVA237 — NVA237 (Glycopyrronioum bromide) as a powder for inhalation in single-dose capsules
  Arms: NVA237
Drug: Placebo — Placebo powder for inhalation in single-dose capsules (matching those for NVA237).
  Arms: Placebo

SUMMARY:
The study serves to determine whether the treatment of patients with stable, symptomatic Chronic Obstructive Pulmonary Disease (COPD) with the investigational drug NVA237 is efficient and safe. The efficacy and safety of the drug will be tested against a placebo treatment. The primary criterion to assess efficacy will be the difference between the serial lung function measurements of patients who have been treated for 12 weeks with NVA237 versus those that have received placebo treatment for 12 weeks. A serial lung function measurement (FEV1 testing) will be conducted and the "area under the curve" will be the measure for the ability to breathe.

ELIGIBILITY:
Inclusion criteria: 1. Patients with stable, symptomatic Chronic Obstructive Pulmonary Disease (COPD) with airflow obstruction of level 2 and 3 according to the current Global initiative for chronic Obstructive Lung Disease (GOLD) strategy (2011). 2. Patients with Forced Expiratory Volume in one second (FEV1) ≥ 30% and <80 % of the predicted normal, and FEV1/FVC < 0.70 when measured 45 min after the inhalation of 84 µg ipratropium bromide.

3. Current or ex-smokers with at least 10 cigarette pack years smoking history.

Exclusion criteria:

1. Patients with a history of long QT syndrome, with a prolonged QTc measured during screening, or patients who have a clinically significant ECG abnormality at screening.
2. History of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases.
3. Pregnant or nursing (lactating) women. Women of childbearing potential unless using an effective method of contraception.
4. Patients who in the judgment of the investigator, would be at potential risk if enrolled into the study.
5. Patients who have a clinically significant concomitant disease at screening, including but not limited to clinically significant laboratory abnormalities, clinically significant renal, cardiovascular, neurological, endocrine, immunological, psychiatric, gastrointestinal, hepatic, or hematological abnormalities, or with uncontrolled diabetes, which could interfere with the assessment of the efficacy and safety of the study treatment.
6. Patients with a body mass index (BMI) of more than 40 kg/m2.
7. Patients contraindicated for treatment with, or having a history of reactions/ hypersensitivity to anticholinergic agents, long and short acting beta-2 agonists, or sympathomimetic amines.
8. Patients with any history of asthma, with onset of symptoms prior to age 40 years, or patients with a high blood eosinophil count during screening.

Other protocol-defnied inclusion/exclusion criteria may apply.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 432 (Actual)
Dates: Start 2012-11; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (51):
- United States (51):
  - Novartis Investigative Site, *See Various Dept.'s*, Arizona
  - Novartis Investigative Site, Chandler, Arizona
  - Novartis Investigative Site, Fresno, California
  - Novartis Investigative Site, Fullerton, California
  - Novartis Investigative Site, Yorba Linda, California
  - Novartis Investigative Site, Boulder, Colorado
  - Novartis Investigative Site, Wheat Ridge, Colorado
  - Novartis Investigative Site, Lynn Haven, Florida
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, Port Orange, Florida
  - Novartis Investigative Site, Winter Park, Florida
  - Novartis Investigative Site, Conyers, Georgia
  - Novartis Investigative Site, River Forest, Illinois
  - Novartis Investigative Site, Skokie, Illinois
  - Novartis Investigative Site, Evansville, Indiana
  - Novartis Investigative Site, Lexington, Kentucky
  - Novartis Investigative Site, Sunset, Louisiana
  - Novartis Investigative Site, Fall River, Massachusetts
  - Novartis Investigative Site, North Dartmouth, Massachusetts
  - Novartis Investigative Site, Minneapolis, Minnesota
  - Novartis Investigative Site, Plymouth, Minnesota
  - Novartis Investigative Site, Saint Charles, Missouri
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Fremont, Nebraska
  - Novartis Investigative Site, Lincoln, Nebraska
  - Novartis Investigative Site, Omaha, Nebraska
  - Novartis Investigative Site, Cherry Hill, New Jersey
  - Novartis Investigative Site, Albuquerque, New Mexico
  - Novartis Investigative Site, Brooklyn, New York
  - Novartis Investigative Site, Great Neck, New York
  - Novartis Investigative Site, Massapequa, New York
  - Novartis Investigative Site, New Windsor, New York
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Charlotte, North Carolina
  - Novartis Investigative Site, Cincinnati, Ohio
  - Novartis Investigative Site, Columbus, Ohio
  - Novartis Investigative Site, Medford, Oregon
  - Novartis Investigative Site, Portland, Oregon
  - Novartis Investigative Site, Langhorne, Pennsylvania
  - Novartis Investigative Site, Pittsburgh, Pennsylvania
  - Novartis Investigative Site, Pottstown, Pennsylvania
  - Novartis Investigative Site, Tipton, Pennsylvania
  - Novartis Investigative Site, East Providence, Rhode Island
  - Novartis Investigative Site, Fort Mill, South Carolina
  - Novartis Investigative Site, Rock Hll, South Carolina
  - Novartis Investigative Site, Denton, Texas
  - Novartis Investigative Site, San Antonio, Texas
  - Novartis Investigative Site, Midvale, Utah
  - Novartis Investigative Site, South Burlington, Vermont
  - Novartis Investigative Site, Richmond, Virginia
  - Novartis Investigative Site, Tacoma, Washington

REFERENCES:
- [Derived] Kerwin E, Siler TM, Korenblat P, White A, Eckert JH, Henley M, Patalano F, D'Andrea P. Efficacy and Safety of Twice-Daily Glycopyrrolate Versus Placebo in Patients With COPD: The GEM2 Study. Chronic Obstr Pulm Dis. 2016 Mar 28;3(2):549-559. doi: 10.15326/jcopdf.3.2.2015.0157. PMID 28848879

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | NVA237 | Placebo
Started | 216 | 216
Full Analysis Set (FAS) | 215 (patients were analyzed according to the treatment to which they were randomized) | 214
Completed | 209 | 205
Not Completed | 7 | 11
Not completed — Lost to Follow-up | 0 | 2
Not completed — Patient/guardian decision | 7 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NVA237 | Placebo | Total
Number analyzed (Participants) | 216 | 216 | 432
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.9 (8.55) | 64.2 (8.41) | 64.1 (8.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88 | 90 | 178
  Male | 128 | 126 | 254

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Standardized Area Under the Curve for Forced Expiratory Volume in One Second Post Dosing
Description: The standardized Area Under the Curve (AUC) for Forced Expiratory Volume in one second (FEV1) post dosing (FEV1 AUC) is measured at week 12 of treatment. Serial lung function measurements are taken at the following time points following dosing at week 12 to calculate the FEV1 AUC: 5 min, 15 min, 1:00 h, 2:00 h, 4:00 h, 6:00 h, 8:00 h, and 11:55 h after the morning dose.
  The primary endpoint was the change from baseline in FEV1 AUC0-12h following the morning dose at Week 12 (defined as the mean FEV1 change from baseline (CFB) over 5 min to 11 h 55 mins divided by 11 h 50 mins). Where the FEV1 AUC is smaller than at baseline, a negative value can occur
Time Frame: Week 12
Population: The full analysis set (FAS): all randomized patients who received at least one dose of trial drug, patients were analyzed according to the treatment they were assigned to at randomization. analyzed participants had values at both baseline and the corresponding time frame, i.e. week 12
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | NVA237 | Placebo
Number analyzed (Participants) | 215 | 213
Liters | 0.115 (0.0153) | -0.008 (0.0153)

2. Secondary Outcome: Change From Baseline in Standardized Area Under the Curve (AUC(0-12h)) for Forced Expiratory Volume in One Second Post Dosing
Description: The standardized Area Under the Curve (AUC) for Forced Expiratory Volume in one second (FEV1) post dosing (FEV1 AUC) is assessed at day 1 of treatment. Serial lung function measurements are taken at the following various time points post dosing at day 1 to calculate the FEV1 AUC: 5 min, 15 min, 1:00 h, 2:00 h, 4:00 h, 6:00 h, 8:00 h, and 11:55 h after the morning dose.
  .The endpoint was the change from baseline (CFB) in FEV1 AUC0-12h following the morning dose at day 1 (defined as the mean FEV1 change from baseline over 5 min to 11 h 55 mins divided by 11 h 50 mins). Where the FEV1 AUC is smaller than at baseline, a negative value can occur.
Time Frame: Day 1
Population: The full analysis set (FAS): all randomized patients who received at least one dose of trial drug, patients were analyzed according to the treatment they were assigned to at randomization. However, for a given time frame, analyzed participants had values at both baseline and the corresponding time frame, i.e. Day 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | NVA237 | Placebo
Number analyzed (Participants) | 215 | 213
Liters | 0.121 (0.0096) | 0.003 (0.0096)

3. Secondary Outcome: Change From Baseline in Standardized Area Under The Curve for Forced Expiratory Volume in One Second for Different Time Spans Post Dosing
Description: The standardized Area Under the Curve (AUC) for Forced Expiratory Volume in one second (FEV1FEV1) is assessed for different time spans (0-4 h, 4-8 h, 8-12 h) within the overall serial measurement post dosing (FEV1 AUCs Time Spans), at day 1 and at week 12 of treatment. Serial lung function measurements are taken at various the following time points post dosing on day 1 and at week 12 to calculate the FEV1 AUC for these different time spans: .5 min, 15 min, 1:00 h, 2:00 h, 4:00 h, 6:00 h, 8:00 h, and 11:55 h after the morning dose.
  The endpoint was the change from baseline (CFB) in FEV1 AUC0-12h following the morning dose at day 1 or week 12, respectively, (defined as the mean FEV1 change from baseline over 5 min to 11 h 55 mins divided by 11 h 50 mins). Where the FEV1 AUC is smaller than at baseline, a negative value can occur.
Time Frame: Day 1 and Week 12
Population: The full analysis set (FAS): all randomized patients who received at least one dose of trial drug, patients were analyzed according to the treatment they were assigned to at randomization. However, for a given time frame, analyzed participants had values at both baseline and the corresponding time frame, i.e. Day 1and Week 12
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | NVA237 | Placebo
Number analyzed (Participants) | 215 | 214
Liters
  Day 1 AUC 0-4h (n=215,213) | 0.154 (0.0088) | 0.014 (0.0088)
  Week 12 AUC 0-4h (n=215,213) | 0.153 (0.0159) | 0.004 (0.0159)
  Day 1 AUC 4-8h (n=213,209) | 0.118 (0.0107) | 0.011 (0.0109)
  Week 12 AUC 4-8h (n=213,209) | 0.107 (0.0159) | 0.000 (0.0158)
  Day 1 AUC 8-12h (n=212,210) | 0.085 (0.0120) | -0.021 (0.0120)
  Week 12 AUC 8-12h (n=212,210) | 0.075 (0.0164) | -0.033 (0.0164)

4. Secondary Outcome: Change From Baseline in Forced Expiratory Volume in One Second at All Individual Timepoints
Description: The Forced Expiratory Volume in one second (FEV1) assessments for all individual time points of the serial measurements on day 1 and at week 12 are analyzed. Time points of the serial lung function measurements are 5 min, 15 min, 1:00 h, 2:00 h, 4:00 h, 6:00 h, 8:00 h, and 11:55 h after the morning dose. The table indicates the percent change from baseline (CFB) in FEV1 and standard deviation in brackets. Where the FEV1 is lower than at baseline, a negative percent value can occur.
Time Frame: Day 1 and week 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | NVA237 | Placebo
Number analyzed (Participants) | 215 | 214
Percent
  FEV1, day 1, 5 min (n=207,202) | 4.9 (8.67) | -0.3 (7.07)
  FEV1, day 1, 15 min (n=209,201) | 9.9 (10.05) | 0.3 (7.62)
  FEV1, day 1, 1 h (n=205,205) | 13.9 (11.98) | 1.2 (9.05)
  FEV1, day 1, 2 h (n=201,205) | 16.0 (14.42) | 2.5 (9.80)
  FEV1, day 1, 4 h (n=199,202) | 12.7 (13.39) | 2.2 (12.63)
  FEV1, day 1, 6h (n=197,197) | 10.3 (13.82) | 2.2 (11.88)
  FEV1, day 1, 8 h (n=200,189) | 8.9 (14.43) | -0.5 (12.42)
  FEV1, day 1, 11 h 55min (n=184,182) | 6.6 (13.44) | -1.7 (14.03)
  FEV1, day 85, -45min (n=184,188) | 6.4 (17.61) | 1.7 (17.95)
  FEV1, day 85, -15min (n=180,185) | 9.6 (18.23) | 2.7 (17.82)
  FEV1, day 85, 5min (n=185,178) | 10.4 (18.78) | 1.8 (17.22)
  FEV1, day 85, 15min (n=186,189) | 12.9 (20.00) | 2.0 (17.08)
  FEV1, day 85, 1h (n=184,187) | 15.8 (20.49) | 1.6 (17.37)
  FEV1, day 85, 2h (n=178,187) | 16.0 (20.83) | 2.4 (18.52)
  FEV1, day 85, 4h (n=179,183) | 12.5 (19.72) | 3.5 (20.25)
  FEV1, day 85, 6h (n=174,172) | 9.8 (18.78) | 2.5 (20.84)
  FEV1, day 85, 8h (n=178,174) | 7.8 (18.18) | 0.2 (18.86)
  FEV1, day 85, 11h 55min (n=171,171) | 7.2 (19.39) | -2.1 (20.07)

5. Secondary Outcome: Mean Trough Forced Expiratory Volume in One Second
Description: Mean trough Forced Expiratory Volume in one second (FEV1) is assessed as the arithmetic mean of two FEV1 measurements, conducted within the last hour of a 24 hour period from a morning dose, either that of day 1 or at week 12 of treatment. The data is reported as the change from baseline (CFB), with the baseline being the arithmetic mean of the two pre-dose measurements (-45 min and -15 min) preceding the serial lung function measurements on Day 1
Time Frame: Day 1 and week 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | NVA237 | Placebo
Number analyzed (Participants) | 213 | 208
Liters
  Day 1 | 0.128 (0.0129) | 0.021 (0.0130)
  Week 12 | 0.123 (0.0166) | 0.038 (0.0166)

6. Secondary Outcome: Change From Baseline in the Health Status Assessed by St. George's Respiratory Questionnaire
Description: The health status, as reported by the patients, is assessed using the St. George's Respiratory Questionnaire (SGRQ). The SGRQ is a 50 item scale assessing symptoms, patient activities and impact of the disease. Scores range from 0 to 100 units, with higher scores indicating more limitations. The assessment is based on total score as well as the percentage of patients with clinically significant improvement at week 12 versus day 1. A clinically meaningful improvement (MCID) in SGRQ is defined as a decrease of 4 or more units of the SGRQ scale in the total score, as compared to baseline (change from baseline).
Time Frame: Week 12
Population: The full analysis set (FAS): all randomized patients who received at least one dose of trial drug, patients were analyzed according to the treatment they were assigned to at randomization. However, for a given time frame, analyzed participants had values at both baseline and the corresponding time frame, i.e. Week 12
Measure: Least Squares Mean (Standard Error); unit: Score
Arm/Group | NVA237 | Placebo
Number analyzed (Participants) | 193 | 194
Score | -6.4 (1.08) | -1.2 (1.06)

7. Secondary Outcome: Breathlessness Assessed by Transition Dyspnea Index
Description: Breathlessness at week 12 is measured using the interviewer-administered Transition Dyspnea Index (TDI). On day 1, breathlessness is assessed by the interviewer-administered Baseline Dyspnea Index (BDI). The change from BDI to TDI is assessed, with the TDI total score ranging from -9 to +9 units of the scale. The lower the score, the more deterioration in severity of dyspnea. Patients are considered to have clinically significant improvement (MCID) with the TDI score change versus BDI being equal to or greater than 1.
Time Frame: Week 12
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Score
Arm/Group | NVA237 | Placebo
Number analyzed (Participants) | 190 | 190
Score | 0.95 (0.280) | 0.48 (0.277)

8. Secondary Outcome: Change From Baseline in Mean Number of Puffs of Rescue Medication Per Day
Description: Patients report the number of puffs of rescue medication (salbutamol / albuterol) using an electronic diary. The use of rescue medication is analyzed as the change from baseline in the mean daily number of puffs used per patient over the 12 weeks treatment period. The baseline is calculated from the run-in epoch prior to randomization (mean number of puffs per day). A negative number indicates a reduction in the mean daily number of puffs of rescue medication.
Time Frame: Baseline and week 12
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Number of puffs
Arm/Group | NVA237 | Placebo
Number analyzed (Participants) | 208 | 201
Number of puffs | -1.33 (0.163) | -0.80 (0.160)

9. Secondary Outcome: Change From Baseline in the Percentage of Days Without Rescue Medication Use
Description: Patients report the number of puffs of rescue medication (salbutamol / albuterol) using an electronic diary. The use of rescue medication is analyzed as the change from baseline in the percentage of days without usage of rescue medication over the 12 weeks treatment period. The baseline is calculated as the percentage of days without usage of rescue medication from during the the run-in epoch prior to randomization.
Time Frame: Baseline and week 12
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: percentage of days
Arm/Group | NVA237 | Placebo
Number analyzed (Participants) | 206 | 198
percentage of days | 11.4 (1.95) | 7.0 (1.97)

10. Secondary Outcome: Change From Baseline in Daily Symptom Scores
Description: Patients are reporting symptoms by using an electronic diary. The electronic diary has 9 symptom questions each morning and each evening. Each question can be answered with one of four pre-defined answers, corresponding to a unit value of 0-3, where 0 stands for the lowest and 3 for the most severe symptom experience. Symptom scores are calculated as the mean of the combined daily symptom scores (combined from morning and evening scores) for each patient over 12 weeks (Day 1 to week 12). The baseline is calculated from the run-in epoch prior to randomization. The change from baseline in the least squares mean daily symptom scores over the 12 week treatment period is provided. Where the mean daily symptom score over the 12 week treatment period is lower than the baseline, the result is negative. A negative result indicates an improvement in COPD symptom severity.
Time Frame: day 1 to week 12
Population: The full analysis set (FAS): all randomized patients who received at least one dose of trial drug, patients were analyzed according to the treatment they were assigned to at randomization. However, for a given time frame, analyzed participants had values at both baseline and the corresponding time frame.
Measure: Least Squares Mean (Standard Error); unit: Score
Arm/Group | NVA237 | Placebo
Number analyzed (Participants) | 208 | 201
Score | -1.09 (0.103) | -0.80 (0.104)

11. Secondary Outcome: Change From Baseline in the Percentage of Nights With "no Nighttime Awakenings"
Description: Patients are reporting symptoms by using an electronic diary. The electronic diary has 9 symptom questions each morning and each evening. One of the symptom questions of the morning questionnaire relates to the number of awakenings due to COPD symptoms during the previous night. The answer with the lowest symptom score is "no waking due to symptoms." A night with "no nighttime awakening" is defined from diary data as any night where the patient did not wake up due to symptoms. The change from baseline in the percentage of nights with "no nighttime awakening" is calculated from the mean percentage of nights with this answer over the 12 week treatment period, with the baseline being The baseline is calculated from the run-in epoch prior to randomization.
Time Frame: Day 1 and week 12
Population: The full analysis set (FAS): all randomized patients who received at least one dose of trial drug. Following the intent-to-treat principle, patients were analyzed according to the treatment they were assigned to at randomization
Measure: Least Squares Mean (Standard Error); unit: Percentage of nights
Arm/Group | NVA237 | Placebo
Number analyzed (Participants) | 208 | 200
Percentage of nights | 13.1 (1.52) | 9.2 (1.54)

12. Secondary Outcome: Change From Baseline in the Percentage of Days With "no Daytime Symptoms"
Description: Patients are reporting symptoms by using an electronic diary. The electronic diary has 9 symptom questions each morning and each evening. Each question can be answered with one of four pre-defined answers, corresponding to a unit value of 0-3, where 0 stands for the lowest and 3 for the most severe symptom experience. A day with "no daytime symptoms" is defined from diary data as any day where the patient has recorded in the evening no cough, no wheeze, no production of sputum, and no feeling of breathlessness (other than when running) during the past approximately 12 hours in the evening questionnaire. The change from baseline in the percentage of days with "no daytime symptoms" is calculated from the mean percentage of days with this answer over the 12 week treatment period, with the baseline being. The baseline is calculated from the run-in epoch prior to randomization.
Time Frame: Day 1 to week 12
Population: as for outcome 11
Measure: Least Squares Mean (Standard Error); unit: Percentage of days
Arm/Group | NVA237 | Placebo
Number analyzed (Participants) | 207 | 195
Percentage of days | 3.6 (1.17) | 2.6 (1.18)

13. Secondary Outcome: Change From Baseline in Percentage of "Days Able to Perform Usual Daily Activities"
Description: Patients are reporting symptoms by using an electronic diary. The electronic diary has 9 symptom questions each morning and each evening. One of the symptom questions of the evening questionnaire relates to the impact of COPD symptoms on the performance of usual daily activities ("Did your respiratory symptoms stop you performing your usual daily activities today"). The answer with the lowest symptom score is "not at all." A "day able to perform usual daily activities" is defined from diary data as any day where the patient was not prevented from performing their usual daily activities due to respiratory symptoms. The change from baseline in the percentage of "days able to perform usual daily activities" is calculated from the mean percentage of days with this answer over the 12 week treatment period, with the baseline beingThe baseline is calculated from the run-in epoch prior to randomization.
Time Frame: Day 1 to week 12
Population: as for outcome 11
Measure: Least Squares Mean (Standard Error); unit: Percentage of days
Arm/Group | NVA237 | Placebo
Number analyzed (Participants) | 207 | 195
Percentage of days | 5.2 (1.61) | 0.9 (1.65)

14. Secondary Outcome: Change From Baseline in Forced Vital Capacity at All Individual Timepoints
Description: The Forced Vital Capacity (FVC)assessments for all individual time points of the serial measurements on day 1 and at week 12 are analyzed. Serial lung function measurements are taken at the following time points following dosing on Day 1 and at week 12: 5 min, 15 min, 1:00 h, 2:00 h, 4:00 h, 6:00 h, 8:00 h, and 11:55 h after the morning dose. For week 12 (day 85), the pre-dose measurements (-45 min and -15 min) and the trough measurements (23:15 h and 23:45 h post-dose) are included. The endpoints are the change from baseline in FVC following the morning dose on Day 1 and at Week 12. Where the FVC at any one timepoint is smaller than at baseline, a negative value can occur.
Time Frame: Day 1 and week 12
Population: as for outcome 11
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | NVA237 | Placebo
Number analyzed (Participants) | 215 | 214
Liters
  FVC, day 1, 5 min (n=214,211) | 0.120 (0.0129) | -0.014 (0.0131)
  FVC, day 1, 15 min (n=214,213) | 0.233 (0.0155) | 0.005 (0.0157)
  FVC, day 1, 1 h (n=215,211) | 0.304 (0.0175) | 0.041 (0.0176)
  FVC, day 1, 2 h (n=211,211) | 0.322 (0.0193) | 0.060 (0.0191)
  FVC, day 1, 4 h (n=209,208) | 0.247 (0.0196) | 0.048 (0.0195)
  FVC, day 1, 6 h (n=208,205) | 0.225 (0.0219) | 0.051 (0.0220)
  FVC, day 1, 8 h (n=209,205) | 0.200 (0.0228) | -0.002 (0.0232)
  FVC, day 1, 11 h 55min (n=203,202) | 0.147 (0.0242) | -0.017 (0.0243)
  FVC, day 85, -45 min (n=207,204) | 0.123 (0.0248) | 0.008 (0.0246)
  FVC, day 85, -15 min (n=208,204) | 0.146 (0.0241) | 0.010 (0.0239)
  FVC, day 85, 5 min (n=214,211) | 0.177 (0.0247) | 0.001 (0.0251)
  FVC, day 85, 15 min (n=214,213) | 0.219 (0.0261) | -0.003 (0.0259)
  FVC, day 85, 1 hr (n=215,211) | 0.267 (0.0261) | 0.010 (0.0260)
  FVC, day 85, 2 hr (n=211,211) | 0.275 (0.0277) | 0.024 (0.0271)
  FVC, day 85, 4 hr (n=209,208) | 0.204 (0.0281) | 0.035 (0.0278)
  FVC, day 85, 6 hr (n=208,205) | 0.185 (0.0278) | 0.016 (0.0278)
  FVC, day 85, 8 hr (n=209,205) | 0.152 (0.0264) | -0.015 (0.0266)
  FVC, day 85, 11 hr 55min (n=203,202) | 0.135 (0.0290) | -0.045 (0.0288)
  FVC, day 85, 23 hr 15min (n=210,204) | 0.207 (0.0289) | 0.066 (0.0284)
  FVC, day 85, 23 hr 45min (n=213,208) | 0.228 (0.0292) | 0.095 (0.0290)

15. Secondary Outcome: Change From Baseline in Mean Trough Forced Vital Capacity
Description: Mean trough Forced Vital Capacity (FVC) is assessed as the arithmetic mean of two FVC measurements, conducted within the last hour of a 24 hours period from a morning dose, either that of day 1 or at week 12 of treatment (23:15 h and 23:45 h assessments). The endpoints are the change from baseline in trough FVC on Day 1 and at Week 12, with the mean of the -45 min and -15 min measurements on Day 1 as the baseline.
Time Frame: Day 1 and week 12
Population: as for outcome 11
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | NVA237 | Placebo
Number analyzed (Participants) | 213 | 208
Liters
  Day 1 | 0.249 (0.0225) | 0.078 (0.0227)
  Week 12 | 0.210 (0.0277) | 0.080 (0.0276)

16. Secondary Outcome: Change From Baseline in Morning and Nighttime Symptom Scores
Description: Patients are reporting morning and nighttime symptoms by using an electronic diary. The electronic diary has 9 symptom questions each morning and each evening. Each question can be answered with one of four pre-defined answers, corresponding to a unit value of 0-3, where 0 stands for the lowest and 3 for the most severe symptom experience. Morning and nighttime symptoms scores for each patient over 12 weeks are reported and analyzed. Symptom scores are calculated as the mean of the symptom scores (morning symptom scores or nighttime symptom scores, respectively) for each patient over 12 weeks (Day 1 to week 12). The baseline is calculated from the run-in epoch prior to randomization. The outcome is calculated as the change from baseline in the morning and nighttime symptom scores, respectively. A negative number indicates a reduction in the symptom severity and is owed to the calculation of the change from baseline.
Time Frame: Day 1 to week 12
Population: as for outcome 11
Measure: Least Squares Mean (Standard Error); unit: Score
Arm/Group | NVA237 | Placebo
Number analyzed (Participants) | 215 | 214
Score
  Daytime total symptom score (n=207,195) | -0.86 (0.097) | -0.61 (0.100)
  Nighttime total symptom score (n=208,200) | -1.03 (0.101) | -0.76 (0.102)

ADVERSE EVENTS:
Arm/Group | NVA237 | Placebo
Serious Adverse Events (participants affected / at risk) | 9/216 | 5/214
Other Adverse Events (participants affected / at risk) | 88/216 | 81/214
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NVA237 (N=216) | Placebo (N=214)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 | 0
ANGINA PECTORIS (Cardiac disorders) | 1 | 0
CELLULITIS (Infections and infestations) | 1 | 0
HERPES SIMPLEX (Infections and infestations) | 1 | 0
OPHTHALMIC HERPES ZOSTER (Infections and infestations) | 1 | 0
PNEUMONIA (Infections and infestations) | 1 | 0
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
METASTATIC SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
SQUAMOUS CELL CARCINOMA OF THE VULVA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 3 | 3
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PULMONARY MASS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PERIPHERAL ARTERY ANEURYSM (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 0.9% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NVA237 (N=216) | Placebo (N=214)
VISION BLURRED (Eye disorders) | 1 | 2
CONSTIPATION (Gastrointestinal disorders) | 1 | 2
DIARRHOEA (Gastrointestinal disorders) | 2 | 3
DRY MOUTH (Gastrointestinal disorders) | 2 | 1
NAUSEA (Gastrointestinal disorders) | 2 | 0
FATIGUE (General disorders) | 1 | 2
OEDEMA PERIPHERAL (General disorders) | 1 | 3
PAIN (General disorders) | 2 | 0
BRONCHITIS (Infections and infestations) | 0 | 4
CANDIDA INFECTION (Infections and infestations) | 3 | 0
CELLULITIS (Infections and infestations) | 2 | 0
GASTROENTERITIS (Infections and infestations) | 2 | 0
GASTROENTERITIS VIRAL (Infections and infestations) | 2 | 3
NASOPHARYNGITIS (Infections and infestations) | 5 | 2
ORAL CANDIDIASIS (Infections and infestations) | 2 | 0
SINUSITIS (Infections and infestations) | 3 | 2
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 7 | 3
URINARY TRACT INFECTION (Infections and infestations) | 3 | 3
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 | 3
ACCIDENTAL OVERDOSE (Injury, poisoning and procedural complications) | 2 | 1
FALL (Injury, poisoning and procedural complications) | 1 | 2
MUSCLE STRAIN (Injury, poisoning and procedural complications) | 1 | 2
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 2 | 1
BLOOD PRESSURE INCREASED (Investigations) | 2 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 | 0
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 2 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 5 | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 2 | 0
DIZZINESS (Nervous system disorders) | 3 | 2
HEADACHE (Nervous system disorders) | 2 | 7
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 43 | 43
COUGH (Respiratory, thoracic and mediastinal disorders) | 6 | 6
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 3 | 3
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 5
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 5 | 1
RESPIRATORY TRACT CONGESTION (Respiratory, thoracic and mediastinal disorders) | 2 | 1
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 3 | 0
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 3
RASH (Skin and subcutaneous tissue disorders) | 1 | 2
HYPERTENSION (Vascular disorders) | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety